CLINICAL TRIAL: NCT03071549
Title: Clinical and Dermoscopic Study Using a Combination of Salicylic and Azaleic Acid Verus Trichloroacetic Acid 25% Peel in Treatment of Mild to Moderate Acne , A Split Face, Double Blinded, Randomised Controlled Trial
Brief Title: Combined Salicylic and Azaleic Acid Verus Trichloroacetic Acid 25% Peel in Treatment of Acne
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rania Abdel hay, Associate professor of dermatology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Dermatology REC 3/2016
Record Dates: First submitted 2017-02-26; First posted 2017-03-07 (Actual); Last update posted 2017-03-07 (Actual); Status verified 2017-03

CONDITIONS: Acne Vulgaris
Keywords: Acne vulgaris; Chemical peeling; Dermoscopy
MeSH Terms: conditions — Acne Vulgaris | interventions — Salicylates

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- combined azaleic and salicylic acids (Active Comparator): Combined azaleic acid 20% with salicylic acid 20% peel every 2 weeks for 4 sessions
  Interventions: Drug: combined azaleic and salicylic acids
- Trichloroacetic acid peel (Active Comparator): Trichloroacetic acid 25% peel every 2 weeks for 4 sessions
  Interventions: Drug: Trichloroacetic acid peel

INTERVENTIONS:
Drug: Trichloroacetic acid peel — Skin degreasing will be performed before every session using acetone. Trichloroacetic acid 25% will be applied on one side of the face.
  Arms: Trichloroacetic acid peel
Drug: combined azaleic and salicylic acids — Skin degreasing will be performed before every session using acetone. Azaleic acid 20% with salicylic acid 20% will be applied to the other side of the face.
  Arms: combined azaleic and salicylic acids

SUMMARY:
Acne patients were included in this randomized controlled trial. Each patient received four treatment sessions two weeks apart. 20% azelaic acid combined with 20% salicylic acid were applied to the one side of the face while 25% trichloroacetic acid was applied to the other side. Evaluation was done by counting number of non-inflammatory and inflammatory lesions before, after two and after four treatment sessions. The dermoscope was used in evaluating the degree of improvement of erythema.

DETAILED DESCRIPTION:
This study included 34 patients with mild and moderate acne vulgaris. The patients were recruited from the dermatology outpatient clinic of Kasr AlAiny hospital.

This study was approved by the Ethical committee of the Faculty of Medicine Cairo University and the Ethical committee of the Dermatology department Cairo University.

After signing an informed consent, patients were subjected to history taking, clinical examination and grading of their acne by global acne grading score, photography, dermoscopic examination and chemical peeling.

Photography:

Patient was photographed from front, lateral and side view before each session and two weeks after the 4th session. All photographs were taken using a digital camera (Nikon AW1, Indonesia) with identical lightening and patient positions.

Dermoscopy:

The cheek was split as four quadrants and photography of dermoscopic figures was taken before every session and two weeks after the 4th session (Using Dermalite DL3N Gen, USA).

Chemical peeling:

Skin degreasing was performed before every session using acetone. Trichloroacetic acid 25% was applied on one side of the face and azaleic acid 20% with salicylic acid 20% to the other side of the face randomly. Randomization was done through a computer-generated random sequence prepared by a statistician; Allocation was concealed in sequentially numbered, sealed, opaque envelopes, and kept by a nurse not involved in the study.

A gauze was used to apply the peel. The gauze was soaked with the peel. The peel was applied uniformly starting from medial to lateral. The peel was left on each side for around 60 seconds. The patients were asked to wash their faces using tape water for neutralization of the peel until the burning sensation is eliminated.

Patients received 4 sessions 2 weeks apart. As a post procedure care, the patients were asked to apply sun screens immediately after the procedure until their next session.

No other topical or systemic treatment was used during sessions. Patients will receive 4 peeling sessions 2 weeks apart.

ELIGIBILITY:
Inclusion Criteria:

* any patients with active acne

Exclusion Criteria:

1. Pregnancy.
2. History of oral herpes simplex virus.
3. History of keloid formation.
4. Associated autoimmune disease (e.g vitiligo, systemic lupus erythematosus).
5. History of past medications in the last six months.
6. Patient unable to perform necessary postoperative care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Change in acne lesions count | 8 weeks
  Change from baseline inflammatory and non-inflammatory lesions count at 2 months

SECONDARY OUTCOMES:
change in acne erythema grading | 2 months
  Change from baseline acne erythema grading using dermoscopy at 2 months

IPD SHARING:
Plan to Share IPD: No